CLINICAL TRIAL: NCT02912065
Title: Tube Feeding Tolerance After Switch to Peptide Based Formula in Children With Developmental Delay: A Retrospective Assessment
Brief Title: Tube Feeding Tolerance After Switch to Peptide Based Formula in Children With Developmental Delay
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 14.08.US.HCN
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Developmental Disabilities; Feeding Disorder
MeSH Terms: conditions — Developmental Disabilities; Feeding and Eating Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective chart review to assess feeding tolerance in children who had been switched from an intact protein formula to a Peptide based formula due to feeding intolerance in a pediatric facility for the developmentally delayed.

DETAILED DESCRIPTION:
Medical records of pediatric patients with enteral feeding intolerance on standard polymeric formulas that were switched to a peptide based formula will be retrospectively analyzed. Data will be collected on caloric intake, ability to meet enteral nutrition goals, incidence of intolerance, and the use of medications to control gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 13 months to < 18 years of age on admission to facility
* Required enteral nutrition to meet 90% or more of their energy needs prior to switch to a Peptide based formula
* Received enteral nutrition with an intact protein formula for a minimum of two weeks prior to a switch to a Peptide based formula
* Have documentation of intolerance to an intact protein formula, followed by a switch in formula received to a Peptide based formula
* Have documentation of an assessment of feeding tolerance following the switch to a Peptide based formula
* Formulas received must be indicated for use in children or adults (not infant formulas).

Exclusion Criteria:

* Recent abdominal surgery, change in tube position/placement (within past 30 days)
* Cow's milk protein allergy
* Any current infections including upper respiratory, viral, gastroenteritis, wound infection.

Ages: 13 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population studied retrospectively will be pediatric patients with developmental delays dependent on enteral nutrition for 90% or more of their nutritional needs and meeting the inclusion/ exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Feeding tolerance after switching to Peptide based formula | up to 30 days post formula switch
  Categorized as no change, tolerance improved, tolerance worsened.

SECONDARY OUTCOMES:
Intake of target feeding volume | up to 30 days post formula switch
  Documentation of feeding volume after switch as "less than," "about the same as," or "more than" feeding volume achieved before switch.
Feeding intolerance parameter(s) identified before switch to Peptide based formula and feeding tolerance parameter(s) improved by switch. | up to 30 days post formula switch
  Intolerance Parameter's: Gagging/retching, vomiting, high residuals, abdominal distention/ gas, stool consistency issues (too hard, too loose).

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Minor, PA-C, Principal Investigator — Childrens Center for Gastroenterology
Locations (1):
- Childrens Center for Gastroenterology, Hollywood, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All data will be presented in manuscript